CLINICAL TRIAL: NCT06691204
Title: Comparison of Adductor Pollicis and Abductor Digiti Minimi Muscles (Thumb Vs. Fifth Digit) As Sites for Neuromuscular Monitoring with Electromyography
Status: Recruiting | Type: Observational
Sponsor: Tamas Vegh, MD (Other)
Responsible Party: Sponsor-Investigator, Tamas Vegh, MD, Head, Division of General, Vascular and Thoracic Anesthesia, University of Debrecen
Organization: University of Debrecen (Other)
Other Study IDs: AITT 2023/7; DE RKEB/IKEB 6656-2023 (Other: Regional and Institutional Ethics Committee University of Debrecen Clinical Center); BM/26645-1/2024 (Other: Ministry of Interior, Research Council Mailing)
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Residual Curarization; Neuromuscular Blockade
Keywords: Electromyography
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the performance of the TetraGraph on two muscle groups: the adductor pollicis and the abductor digiti minimi. Theese muscles are located on the arms. Key time points for assessment will include the onset of neuromuscular blockade and the recovery from rocuronium blockade using sugammadex.

DETAILED DESCRIPTION:
Introduction Residual neuromuscular blockade is a common occurrence in the post-anesthesia care unit (PACU) when neuromuscular blocking agents (NMBAs) have been used in the operating room. The only method of reliably detecting residual neuromuscular blockade is through the use of quantitative neuromuscular monitors. Unfortunately, several barriers exist that have prevented the widespread use of these devices. For instance, there is a paucity of quantitative neuromuscular monitors commercially available. Also, two modalities of quantitative monitoring, kinemyography and acceleromyography, rely on movement of the muscles of interest, a characteristic frequently compromised during patient positioning for surgical procedures in which the patient's arms are secured under surgical drapes (laparoscopic, bariatric, robotic, spine, and neurosurgical procedures) or in uncooperative awake patients in the PACU or intensive care unit (ICU). The aim of this investigation is to determine the different muscle sensitivities to NMBA and reversal agents by comparing responses at two different monitoring sites as measured with a new quantitative monitor. EMG measures electrical activity within the muscle following peripheral nerve stimulation and is unaffected by involuntary patient motion or by restricted muscle movements from surgical positioning. We plan to compare measurements obtained with two TetraGraph devices, one monitoring the adductor pollicis (thumb) muscle and the other monitoring adductor digiti minimi (5th digit) muscle, during onset, maintenance, and recovery of neuromuscular blockade. This will include monitoring every 20 sec for onset of blockade (defined as time from Train-of-Four ratio, TOFR=1.0 until Train-of-four count, TOFC=0) following rocuronium administration, during maintenance of neuromuscular block as required by surgical conditions, and following reversal administration until adequate recovery is documented (train-of-four ratio, TOFR ≥0.9).

Medication of the patient, surgical procedure

Upon entering the operating room, all patients underwent monitoring using electrocardiograms, noninvasive blood pressure measurements, and pulse oximetry. An intravenous catheter was inserted into either the forearm or the dorsal vein. Anesthesia was initiated with intravenous fentanyl (2.0 mg/kg) and propofol (1.5 to 2.5 mg/kg) and was maintained using sevoflurane (end-tidal concentration of 1.0 to 1.3%) in an air-oxygen mixture, with additional fentanyl given as needed. Before tracheal intubation, the patients were manually ventilated with 100% oxygen via facemask. Oxygen saturation was kept above 96%, and normocapnia was maintained. A forced air warming system (Bair Hugger, Arizant Healthcare Inc., Eden Prairie, Minnesota, USA) was used to keep the body temperature at or above 36°C. Intraoperative hypotension was treated with ephedrine, norepinephrine, or a fluid bolus, according to clinical indications. Ondansetron 4mg IV was routinely administered to prevent postoperative nausea and vomiting.

Neuromuscular Management Before the induction of anesthesia, after appropriate skin cleaning, single-use surface TetraGraph electrodes were placed over the ulnar nerve and thumb to assess the adductor pollicis response on one hand, and over the ulnar nerve and fifth digit to assess the abductor digiti minimi response on the other hand. Following the induction of anesthesia, train-of-four (TOF) stimulation was applied to both muscle groups at a frequency of 2 Hz for 1.5 seconds every 15 seconds, after the automated calibration of supramaximal current and responses. Once stable baseline TOF responses were established, all patients received 0.6 mg/kg of rocuronium intravenously. Measurements were taken every five minutes during the intraoperative period until the administration of sugammadex. After that, we monitored the spontaneous recovery of the rocuronium-induced neuromuscular block until three consecutive TOF counts of 2 (TOFC2) were observed at both monitoring sites. Additional doses of rocuronium (0.1-0.2 mg/kg) were administered as necessary to maintain a Train of Four (TOF) count of ≤2. At the end of the surgery, sugammadex was given at a dose of 2 mg/kg. After administering sugammadex, measurements were taken every 20 seconds until the patient was extubated. Following the measurements obtained with both devices at the specified intervals, and once the TOF ratio exceeded 0.9, the devices were disconnected, and the patients continued along the standard recovery pathway.

Rescue medication After pharyngoscopy, rescue medication is given if necessary, i.e. below 90% TOF, depending on the type of muscle relaxant used. If an aminosteroid muscle relaxant is used, the patient is given 2 mg/kg sugammadex, while if a benzylisoquinoline muscle relaxant is used, 0.05 mg/kg neostigmine and 0.015 mg/kg atropine are administrated to antagonise the drug effect.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Patients willing to participate and provide an informed consent
* Patients undergoing elective surgical procedures that require use of NMBA agents (rocuronium) administered intraoperatively.

Exclusion Criteria:

* Patients with disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis.
* Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents, i.e., severe renal impairment or end-stage liver disease.
* Patients having surgery that would involve prepping the arm into the sterile field.
* Patients receiving a rapid sequence induction.
* Patients allergic to rocuronium or sugammadex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive a muscle relaxant (rocuronium bromide) for their operation to aid intubation and surgical exploration.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The rate of recovery following sugammadex administration as recorded simultaneously from the hand (adductor pollicis) and fifth digit (abductor digiti minimi) muscles | depends on the depth of the neuromuscular block, a maximum of about 20 minutes
  the time in seconds between the administration of the suggamedex and TOF 100%.

SECONDARY OUTCOMES:
The incidence of postoperative residual weakness | one hour after extubation
  The secondary endpoint is the incidence of postoperative residual weakness at the time of extubation at a center that predominately utilizes quantitative monitoring (defined as TOFR <0.90).

CONTACTS AND LOCATIONS:
Overall Officials: Béla Fülesdi, MD, Phd, DSc, Study Director — Department of Anesthesiology and Intensive Care University of Debrecen
Locations (2):
- Hungary (2):
  - University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar
  - University of Debrecen, Debrecen, Hajdú-Bihar 4008, Debrecen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nemes R, Fulesdi B, Pongracz A, Asztalos L, Szabo-Maak Z, Lengyel S, Tassonyi E. Impact of reversal strategies on the incidence of postoperative residual paralysis after rocuronium relaxation without neuromuscular monitoring: A partially randomised placebo controlled trial. Eur J Anaesthesiol. 2017 Sep;34(9):609-616. doi: 10.1097/EJA.0000000000000585. PMID 28030444
- [Background] Naguib M, Brull SJ, Kopman AF, Hunter JM, Fulesdi B, Arkes HR, Elstein A, Todd MM, Johnson KB. Consensus Statement on Perioperative Use of Neuromuscular Monitoring. Anesth Analg. 2018 Jul;127(1):71-80. doi: 10.1213/ANE.0000000000002670. PMID 29200077
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Blobner M, Hunter JM, Meistelman C, Hoeft A, Hollmann MW, Kirmeier E, Lewald H, Ulm K. Use of a train-of-four ratio of 0.95 versus 0.9 for tracheal extubation: an exploratory analysis of POPULAR data. Br J Anaesth. 2020 Jan;124(1):63-72. doi: 10.1016/j.bja.2019.08.023. Epub 2019 Oct 10. PMID 31607388
- [Background] Kirmeier E, Eriksson LI, Lewald H, Jonsson Fagerlund M, Hoeft A, Hollmann M, Meistelman C, Hunter JM, Ulm K, Blobner M; POPULAR Contributors. Post-anaesthesia pulmonary complications after use of muscle relaxants (POPULAR): a multicentre, prospective observational study. Lancet Respir Med. 2019 Feb;7(2):129-140. doi: 10.1016/S2213-2600(18)30294-7. Epub 2018 Sep 14. PMID 30224322
- [Background] Herbstreit F, Peters J, Eikermann M. Impaired upper airway integrity by residual neuromuscular blockade: increased airway collapsibility and blunted genioglossus muscle activity in response to negative pharyngeal pressure. Anesthesiology. 2009 Jun;110(6):1253-60. doi: 10.1097/ALN.0b013e31819faa71. PMID 19417617
- [Background] Eikermann M, Vogt FM, Herbstreit F, Vahid-Dastgerdi M, Zenge MO, Ochterbeck C, de Greiff A, Peters J. The predisposition to inspiratory upper airway collapse during partial neuromuscular blockade. Am J Respir Crit Care Med. 2007 Jan 1;175(1):9-15. doi: 10.1164/rccm.200512-1862OC. Epub 2006 Oct 5. PMID 17023729
- [Background] Arbous MS, Meursing AE, van Kleef JW, de Lange JJ, Spoormans HH, Touw P, Werner FM, Grobbee DE. Impact of anesthesia management characteristics on severe morbidity and mortality. Anesthesiology. 2005 Feb;102(2):257-68; quiz 491-2. doi: 10.1097/00000542-200502000-00005. PMID 15681938
- [Background] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Background] Ledowski T, Hillyard S, O'Dea B, Archer R, Vilas-Boas F, Kyle B. Introduction of sugammadex as standard reversal agent: Impact on the incidence of residual neuromuscular blockade and postoperative patient outcome. Indian J Anaesth. 2013 Jan;57(1):46-51. doi: 10.4103/0019-5049.108562. PMID 23716766
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/8394051/